CLINICAL TRIAL: NCT02483104
Title: A Phase 1 Study of Veliparib in Combination With Carboplatin And Weekly Paclitaxel in Japanese Subjects With Ovarian Cancer
Brief Title: Veliparib in Combination With Carboplatin And Weekly Paclitaxel in Japanese Subjects With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-488
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2016-08

CONDITIONS: Ovarian Cancer
Keywords: ABT-888; BRCA; Primary peritoneal cancer; carboplatin; Fallopian tube; Poly (ADP-ribose) polymerase (PARP); paclitaxel; Ovarian cancer; veliparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — veliparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- veliparib (ABT-888) (Experimental)
  Interventions: Drug: veliparib; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: veliparib — Veliparib will be given orally, twice daily on Days 1-21, every 21 days.
  Other Names: ABT-888
Drug: carboplatin — Carboplatin will be administered on Day 1 of each cycle, intravenously.
  Other Names: paraplatin
Drug: paclitaxel — Paclitaxel will be administered on Days 1, 8, 15 of each cycle, intravenously.
  Other Names: taxol

SUMMARY:
This is a Phase 1, open-label, multicenter, dose escalation study evaluating the tolerability, safety, pharmacokinetics and preliminary efficacy of veliparib in combination with carboplatin and weekly paclitaxel in Japanese subjects with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed epithelial ovarian, fallopian tube or primary peritoneal carcinoma the International Federation of Gynecology and Obstetrics (FIGO) Stage IC - IV with either optimal (< 1 cm residual disease) or suboptimal residual disease.

Participants must be newly diagnosed, chemotherapy-naïve, and entered between 1 and 12 weeks after initial cytoreductive surgery.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.

Adequate organ and marrow function.

Ability to swallow and retain oral medication, and no uncontrolled emesis.

Women of childbearing potential (except vasectomized partner of female subjects) must agree to use adequate contraception prior to study entry, for the duration of study participation and up to 3 months following completion of therapy. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to the study entry. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

A history of another invasive cancer within the past 3 years, except non-melanoma skin cancer or in situ malignancies that are considered cured by the investigator (e.g., cervical cancer in situ, in situ carcinoma of the bladder, or breast carcinoma in situ).

Participants who received prior radiotherapy to any portion of the abdominal cavity or pelvis.

Participants who received prior chemotherapy for any abdominal or pelvic tumor.

Any investigational agents less than 4 weeks prior to study enrollment.

Any anti-cancer Chinese medicine/herbal remedies within 14 days prior to study enrollment.

Known history of allergic reaction to Cremophor-paclitaxel, carboplatin, Azo Colourant Tartrazine (also known as FD&C Yellow 5 or E102), Azo Colourant Orange Yellow-S (also known as FD&C Yellow 6 or E110) or known contraindications to any study supplied drug.

Patients with history or evidence upon physical examination of central nervous system disease, including primary brain tumor, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months of the first date of treatment on this study.

Prior therapy with a Poly-(ADP-ribose)-Polymerase (PARP) inhibitor.

Subject has a clinically significant uncontrolled condition(s), including but not limited to:

* Uncontrolled seizure disorder, or focal or generalized seizure within the last 12 months;
* Active infection that requires parenteral antibiotics;
* Known active hepatitis B or hepatitis C with abnormal liver function test or organ dysfunction;
* Symptomatic congestive heart failure; unstable angina pectoris; serious ventricular cardiac arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication (this does not include asymptomatic atrial fibrillation with controlled ventricular rate); or myocardial infarction within the last 6 months;
* Uncontrolled hypertension (sustained systolic blood pressure > 150 mmHg or diastolic pressure > 100 mmHg despite optimal medical management);
* Bowel obstruction or gastric outlet obstruction;
* Psychiatric illness/social situations that would limit compliance with study requirements;
* Any medical condition which in the opinion of the Investigator places the subject at an unacceptably high risk for toxicities.

Pregnant or lactating.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicities | During the first cycle (21 days) of veliparib administration

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 5 months
  Collect all adverse events at each visit and assess according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03
Preliminary tumor response | Participants will be evaluated for 5 months.
  According to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Maximum observed plasma concentration (Cmax) of Veliparib | For 24 hours following veliparib dosing.
  Maximum observed concentration, occurring at Tmax
The time to Cmax (peak time, Tmax) of Veliparib | For 24 hours following veliparib dosing.
  The time at which maximum plasma concentration (Cmax) is observed.
The area under the plasma concentration-time curve (AUC) of Veliparib | For 24 hours following veliparib dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Hashiba, BS, Study Director — AbbVie
Locations (3):
- Japan (3):
  - Site Reference ID/Investigator# 128815, Kurume-shi,Fukuoka
  - Site Reference ID/Investigator# 128997, Morioka
  - Site Reference ID/Investigator# 128058, Nagaizumi-cho

REFERENCES:
- [Result] Nishio S, Takekuma M, Takeuchi S, Kawano K, Tsuda N, Tasaki K, Takahashi N, Abe M, Tanaka A, Nagasawa T, Shoji T, Xiong H, Nuthalapati S, Leahy T, Hashiba H, Kiriyama T, Komarnitsky P, Hirashima Y, Ushijima K. Phase 1 study of veliparib with carboplatin and weekly paclitaxel in Japanese patients with newly diagnosed ovarian cancer. Cancer Sci. 2017 Nov;108(11):2213-2220. doi: 10.1111/cas.13381. Epub 2017 Sep 18. PMID 28837250